CLINICAL TRIAL: NCT03388060
Title: Shockwave Lithotripsy (SWL) Versus Oral Dissolution Therapy (ODT) Versus Combined SWL And ODT For Radiolucent Renal Stone Randomised Controlled Trial
Brief Title: (SWL) Versus (ODT) Versus Combined SWL And ODT For Radiolucent Stone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelbaset, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RL STONE
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Urologic Diseases; Stone, Urinary; Stone, Kidney; ESWL; Radiolucent Calculus of Urinary Tract; Dissolution
Keywords: Oral Dissolution Therapy; Kidney stone; ESWL
MeSH Terms: conditions — Urologic Diseases; Urinary Calculi; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound guided SWL (Active Comparator): ultrasound guided SWL for Radiolucent stone
  Interventions: Procedure: Ultrasound guided SWL
- Dissolution therapy (Active Comparator): Dissolution therapy for Radiolucent stone
  Interventions: Procedure: Dissolution therapy
- Combined ultrasound guided SWL and dissolution therapy (Active Comparator): Combined treatment for Radiolucent stone.
  Interventions: Procedure: Combined ultrasound guided SWL and dissolution therapy

INTERVENTIONS:
Procedure: Ultrasound guided SWL — Ultrasound guided SWL for radiolucent renal stone
  Arms: Ultrasound guided SWL
Procedure: Dissolution therapy — Alkalinization dissolution therapy for radiolucent renal stone
  Arms: Dissolution therapy
Procedure: Combined ultrasound guided SWL and dissolution therapy — Combined ultrasound guided SWL and alkalinization dissolution therapy for radiolucent renal stone
  Arms: Combined ultrasound guided SWL and dissolution therapy

SUMMARY:
compare the efficacy of of ultrasound guided SWL versus dissolution therapy versus combined SWL and dissolution therapy in management of 1 - 2.5 cm renal stones.

DETAILED DESCRIPTION:
Urolithiasis is a common morbidity worldwide, affecting 10% to 15% of the population in Europe and North America. A higher prevalence of stone disease is found in hot or dry areas, including 20% to 25% in the Middle East. Radiolucent stones are mostly uric acid (UA) calculi, which varies geographically with worldwide incidence ranges from 5 to 40% and about 7- 10 percent of all calculi. Other rare radiolucent stones include xanthine and 2,8-dihydroxyadenine calculi.

The main etiologic factors for the development of uric acid nephrolithiasis are low urinary pH, hyperuricosuria, and low urinary volume. Practically, all of those who form uric acid stones have persistently low urinary pH, and most excrete normal amounts of uric acid. This suggests the potential importance of urinary pH manipulation in dissolving UA stones. Dissolution therapy for UA calculi is based on hydration and raising the urinary pH. European guidelines recommended that urine pH should be increased to a level above 6. The early published papers discussed the efficacy of oral chemo-dissolution therapy reporting high success rates. Since that era, there have been only a few publications, with widely variable results (15-80% complete dissolution rate).

Retrograde intrarenal surgery (RIRS), shockwave lithotripsy (SWL), and percutaneous nephrolithotomy (PCNL) are the three main non-medical modalities for treating medium-sized renal stones. Resorlu et al., retrospectively compare the outcomes of SWL, PNL, and RSIS for 10-20 mm radiolucent renal calculi of 437 patients and concluded that success rates "defined as stone-free status or asymptomatic insignificant residual fragments <3 mm." were 66.5, 91.4, and 87 % for SWL, PNL, and RIRS (p<0.001). in a prospective randomized of 135 patient with 1 to 2 cm radiolucent lower calyceal renal calculi, the 3-month stone-free rate of SWL, RIRS and miniperc was 73.8%, 86.1% and 95.1%, respectively (p =0.01).

Comparing the medical in the form of dissolution therapy versus non-medical in the form of SWL, Elderwy et al, in a prospective study on 87 children with radiolucent renal calculi with length less than 25 mm and a normal upper urinary tract or grade I HN, found that stone-free rate was 72.9% for dissolution therapy vs 82.1% after a single session of shock wave lithotripsy (p = 0.314).

Dissolution success is related to stone size as well as compliance. Larger stones demand longer therapy, and in these cases SWL may increase treatment efficacy by increasing stone surface area. So when Mokhless et al., use combined extracorporeal shock wave lithotripsy and dissolution therapy in radiolucent stone 12-65 mm in the largest diameter, stone-free rate of 100% was achieved in all 24 children after 3 months.9 To the best of our knowledge, there is no controlled trial comparing the efficacy of ultrasound guided SWL versus dissolution therapy versus combined SWL and dissolution therapy in management of 1 - 2.5 cm single renal stone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with 1-2.5 cm renal stones.
* Normal Serum creatinine
* Radiolucent stone by X-ray

Exclusion Criteria:

* Pregnancy.
* Bleeding diatheses.
* Patients with a pacemaker.
* Uncontrolled UTIs.
* Severe skeletal malformations.
* Severe obesity which prevent targeting of the stone; BMI (40 or more).
* Arterial aneurysm in the vicinity of the stone.
* Anatomical obstruction distal to the stone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Stone free rate | 3 months
  Free renal units from stones

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Sheir, MD, Study Chair — Shock wave unit chief - Urology and nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt